CLINICAL TRIAL: NCT06342661
Title: Study On the Expression Level and Clinical Significance of VISTA in Patients With Vascular Cognitive Impairment
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022IIT205
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Cerebrovascular Disease Small Vessel
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control
  Interventions: Diagnostic Test: Neuropsychological testing
- Case
  Interventions: Diagnostic Test: Neuropsychological testing

INTERVENTIONS:
Diagnostic Test: Neuropsychological testing — The primary outcomes were Mini-Mental State Examination and Montreal Cognitive Assessment scores for screening of cognitive decline, which are recommended by NINDS-AIREN. The secondary outcomes included the performance in five cognition domains: (1) verbal memory, Hopkins Verbal Learning Test ; (2) visual-spatial ability, Clock Drawing test; (3) executive function, Trail Making test (TMT) (B time); (4) attention, TMT (A time); and (5) language tests, Boston Naming test2 (BNT-2)

SUMMARY:
1. Explore the expression level of immune checkpoint VISTA in peripheral blood and cerebrospinal fluid of patients with cardiovascular risk factors; 2. Discuss the correlation between different risk factors (mainly hypertension, diabetes, smoking, hyperlipidemia, hyperhomocysteinemia, etc.) and the expression level of immune checkpoint VISTA in peripheral blood and cerebrospinal fluid of patients with cerebrovascular diseases and immune-inflammatory related diseases of the nervous system; 3. Explore the correlation between different immune inflammatory factors (IL1, IL6, IL10, INFγ, TNFα) and the expression level of immune checkpoint VISTA in peripheral blood and cerebrospinal fluid of patients; 4. Track and explore the dynamic changes of immune checkpoint VISTA in peripheral blood and cerebrospinal fluid of patients with cardiovascular risk factors in 3 months, 1 year, 3 years, and 5 years.

DETAILED DESCRIPTION:
The prospective observational study design was adopted to screen patients with cardiovascular risk factors who visited the Department of Neurology in the First Hospital of Harbin Medical University since November 2022. The patients mainly categorize into two groups: without cognitive impairment (control) and with cognitive impairment (VCI).. General information, imaging, functional assessment, immune checkpoint VISTA in peripheral blood and cerebrospinal fluid, and blood-related indicators were collected. Some patients who could cooperate were followed up for 3-5 years. By analyzing the correlation between the content of immune checkpoint VISTA in peripheral blood and cerebrospinal fluid, disease risk factors, imaging, functional scores and blood indicators, the relationship between immune checkpoints and nervous system diseases was better understood.

ELIGIBILITY:
Inclusion Criteria:

1. The study included 100 subjects, including 50 patients with VCI and 50 normal controls. The diagnosis of VCI was based on the diagnostic criteria for psychiatric disorders in the fifth revised edition of the "Diagnostic and Statistical Manual of Mental Disorders" of the American Psychiatric Association;
2. All relevant examination and cognitive testing work in this study obtained informed consent from the subjects and their families.

Exclusion Criteria:

1. In line with the exclusion criteria for VCI diagnosis in the "Chinese guidelines for the treatment of vascular cognitive impairment 2019"; complicated with autoimmune diseases, blood diseases, malignant tumors, heart, liver, and kidney dysfunction, infectious diseases, family genetic diseases, recent acute or chronic inflammatory diseases, myocardial infarction, etc.; taking antibiotics, steroids, immunosuppressants before the trial; having a history of cranial trauma or surgery.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively enrolled consecutive patients with cardiovascular risk factors from the First Affiliated Hospital of Harbin Medical University.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Patient characteristics | 2023.03.01-2028.11.30
VISTA expression in PBMCs in the VCI and control groups | 2023.03.01-2028.11.30

CONTACTS AND LOCATIONS:
Overall Officials: 2023.03.01-2028.11.30 Chi, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China